CLINICAL TRIAL: NCT05952596
Title: A Single-center, Randomized, Active-controlled, Parallel-group, Double-blind, Phase I Clinical Trial to Evaluate Safety and Immunogenicity of Hexavalent Vaccine (APV006) in Healthy Adults
Brief Title: A Study to Evaluate Safety and Immunogenicity of APV006 in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LG-VGCL001
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Hepatitis B; Haemophilus Influenzae Type b Infection
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Hepatitis B; Haemophilus Infections

STUDY DESIGN:
Intervention Model Description: active-controlled model
Who Masked: Participant, Investigator
Masking Description: The study pharmacist and study staff who administer the investigational vaccine (e.g., medication nurse) will not be blinded in this study since a control vaccine that can be visually distinguished from the study vaccine will be used. The study staff including the investigator will remain blinded, except the unblinded staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): DTaP-HepB-IPV-Hib vaccine
  Interventions: Biological: DTaP-HepB-IPV-Hib vaccine
- Control group (Active Comparator): DTaP-HepB-IPV-Hib vaccine
  Interventions: Biological: DTaP-HepB-IPV-Hib vaccine

INTERVENTIONS:
Biological: DTaP-HepB-IPV-Hib vaccine — Hexavalent vaccine (DTaP-HepB-IPV-Hib vaccine: Diphtheria-Tetanus-Acelluar Pertussis-Hepatitis B-Sabin Inactivated Poliovirus-Haemophilus influenzae type b vaccine)
  Arms: Test group
Biological: DTaP-HepB-IPV-Hib vaccine — Hexavalent vaccine (DTaP-HepB-IPV-Hib vaccine: Diphtheria-Tetanus-Acellular Pertussis-Hepatitis B-poliomyelitis(inactived)-Haemophilus influenzae type b vaccine)
  Arms: Control group

SUMMARY:
This is a single-center, randomized, active-controlled, parallel-design, double-blind, phase I study to evaluate the safety and immunogenicity of a single dose of APV006 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults aged 19 - 55 on Visit 1
* Those without clinically significant abnormalities on the screening test on Visit 1
* Those with a confirmed BMI of 18.5 kg/m2 to less than 30 kg/m2 on Visit 1
* Those who have heard a detailed explanation of the study and whose written consent to participate in the study was given voluntarily by themselves or their legal representatives

Exclusion Criteria:

* Those who participated in other studies and took investigational products/ investigational vaccines within 6 months from Visit 1
* Those who took tetanus toxoid (TT), tetanus-diphtheria (Td), tetanus-reduced diphtheria-acellular pertussis (Tdap) vaccine for adults, or other vaccines containing tetanus-diphtheria for adults within 5 years from Visit 1
* Those who were vaccinated within 4 weeks from Visit 1 or who plan to receive vaccines other than the investigational vaccine from the participation in this study to Visit 5
* Have had diphtheria, tetanus, pertussis, hepatitis B, polio, or invasive diseases caused by Haemophilus influenzae type b

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-07-17 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with immediate reactions | For 30 minutes after the vaccination
  Immediate reactions after vaccination with the study vaccine mean all the signs and symptoms occurring within 30 minutes after the vaccination.
Number of subjects with solicited adverse events | For 7 days after the vaccination [Day 1-8]
  Solicited adverse events are classified into the local(pain, tenderness, erythema/redness, induration/swelling, pruritus) and systemic(fever, fatigue, chills/shivering, myalgia, headache, arthralgia, decreased appetite, diarrhea, nausea/vomiting, hypersensitivity) signs and symptoms.
Number of subjects with unsolicited adverse events | For 28 days (+7 days of window period) after the vaccination [Day 1-29]
  Unsolicited adverse events mean all the adverse events excluding the solicited adverse events that occur after the ICF is obtained until 28 days after vaccination.
Number of subjects with serious adverse events | For 181 days (+7 days of window period) after the vaccination [Day 1-181]
  serious adverse events that occur after the ICF is obtained until 6 months after vaccination.

SECONDARY OUTCOMES:
Proportions of the subjects who meet seroprotection/vaccine-response to each antigen and the subjects who have shown seroconversion 28 days post-vaccination with the study vaccine (Day 29) compared to pre-vaccination. | Day 29 (+7 days window period)
  Immunogenicity of each components (antibodies against Diphtheria, Tetanus, Acellular Pertussis, Polio, Hepatitis B, and Haemophilus influenzae type b)
Proportion of the subjects who meet one of the following regarding anti-PT, anti-FHA, and anti-PRN | Day 29 (+7 days window period)
  ①If the antibody concentration is < 4 X LLOQ before the administration of the investigational vaccine: The antibody concentration is ≥ 4 X LLOQ 29 days after the administration of the investigational vaccine
  ②If the antibody concentration is ≥ 4 X LLOQ before the administration of the investigational vaccine: The antibody concentration 29 days after the administration of the investigational vaccine is ≥ the antibody concentration before the administration
GMC or GMT values for each antigen prior to and 28 days post-vaccination with the study vaccine (Day 29) | Day 29 (+7 days window period)
  Immunogenicity of each components (antibodies against Diphtheria, Tetanus, Acelluar Pertussis, Polio, Hepatitis B, and Haemophilus influenzae type b

CONTACTS AND LOCATIONS:
Overall Officials: Nam Joong Kim, Principal Investigator — Seoul National University College of Medicine

IPD SHARING:
Plan to Share IPD: No